CLINICAL TRIAL: NCT04316949
Title: Predictors of Respiratory Failure Requiring ICU Admission Among Hospitalized Patients With SARS-Cov-2 Infection
Brief Title: Predictors of Respiratory Failure in SARS-Cov-2 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Michele Bartoletti, Assistant Professor, University of Bologna
Other Study IDs: PREDI-CO
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV-2 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation cohort: Derivation cohort: Italian retrospective cohort of all consecutive hospitalized patients with SARS-CoV-2 pneumonia in the participating centers, from February 20 to March 19 2020.
  .
- Validation cohort: Validation cohort: European and non-European retrospective cohort of all consecutive hospitalized patients with SARS-CoV-2 pneumonia in the participating centers, from March 19 to April 18 2020.

SUMMARY:
The emergence of SARS-CoV-2 is currently engaging and consuming most of resources of efficient healthcare systems in Europe, and several hospitals are currently experiencing a shortage of ICU beds for critically-ill patients with SARS-CoV-2 pneumonia.

A risk stratification based on clinical, radiological and laboratory parameters seems necessary in order to better identify those patients who may need ICU admission and/or those who may benefit from a prompt antiviral therapy

DETAILED DESCRIPTION:
The study will compared patients with and without respiratory failure in order to find risk factors for need for ICU admission. A simple score based on risk factors will be created from a multicenter Italian cohort and validated in a multicenter international cohort.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with microbiologically confirmed diagnosis of SARS-CoV-2 infection
* Age > 17 years

Exclusion Criteria:

* Invasive mechanical ventilation within 12 hours from hospital admission

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study will include all consecutive hospitalized patients with microbiologically confirmed diagnosis of SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory failure | 14 days
  Composite of ICU admission or SpO2<92% with 100% FiO2 of oxygen treatment (reservoir mask or CPAP or NIV), respiratory rate >30 bpm, respiratory distress

SECONDARY OUTCOMES:
Occurence of bacterial superinfection | 14 days
  Incidence of bacterial superinfection among ventilated patients with SARS-CoV-2 pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna - Department of Medical and Surgical Sciences, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Participant from other centers may request to analyze the registry for other purposes upon IRB and study group approval

REFERENCES:
- [Derived] Bartoletti M, Giannella M, Scudeller L, Tedeschi S, Rinaldi M, Bussini L, Fornaro G, Pascale R, Pancaldi L, Pasquini Z, Trapani F, Badia L, Campoli C, Tadolini M, Attard L, Puoti M, Merli M, Mussini C, Menozzi M, Meschiari M, Codeluppi M, Barchiesi F, Cristini F, Saracino A, Licci A, Rapuano S, Tonetti T, Gaibani P, Ranieri VM, Viale P; PREDICO study group. Development and validation of a prediction model for severe respiratory failure in hospitalized patients with SARS-CoV-2 infection: a multicentre cohort study (PREDI-CO study). Clin Microbiol Infect. 2020 Nov;26(11):1545-1553. doi: 10.1016/j.cmi.2020.08.003. Epub 2020 Aug 8. PMID 32781244